CLINICAL TRIAL: NCT06490055
Title: Predicting the Efficacy of Paclitaxel Plus Ramucirumab in Advanced Gastric Cancer.
Brief Title: Predicting the Efficacy in Advanced Gastric Cancer.
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/SLCGC
Record Dates: First submitted 2024-06-21; First posted 2024-07-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer; Chemotherapy Effect; Paclitaxel; Ramucirumab
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; Ramucirumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Blood sample before second-line chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric cancer chemotherapy responders received second-line chemotherapy: Responders according to the response evaluation criteria in solid tumors (RECIST).
  A panel of microRNA, whose expression level is tested exosomal microRNA from blood sample before second-line chemotherapy with reverse transcriptase quantitative polymerase chain reaction (RT-qPCR)
  Interventions: Drug: Paclitaxel
- Gastric cancer chemotherapy non-responders received second-line chemotherapy: Non-responders according to the response evaluation criteria in solid tumors (RECIST).
  A panel of microRNA, whose expression level is tested exosomal microRNA from blood sample before second-line chemotherapy with reverse transcriptase quantitative polymerase chain reaction (RT-qPCR)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Gastric cancer second-line Chemotherapy (paclitaxel plus ramucirumab)
  Other Names: Ramucirumab

SUMMARY:
With advances in chemotherapy for gastric cancer, it is important to identify patients who will respond effectively to specific therapies. This longitudinal study aimed to establish a liquid-biopsy assay that can predict response to ramucirumab plus paclitaxel therapy in patients with advanced gastric cancer.

DETAILED DESCRIPTION:
The combination of paclitaxel and ramucirumab is a potent standard second-line therapy for patients with advanced gastric cancer, but approximately 30% of patients do not respond to treatment. Failure to respond to second-line therapy can lead not only to disease progression, but also to deterioration of the patient's health and loss of the opportunity to receive other treatments that originally had the potential to be curative. This study aims to predict the efficacy of second-line treatment (paclitaxel plus ramucirumab) in patients with gastric cancer using liquid biopsies (small RNA). Prediction using pre-treatment blood may allow patients who do not respond to treatment to choose other treatment options. This study aims to establish a tool that will enable noninvasive pre-treatment selection, which could lead to personalized treatment.

ELIGIBILITY:
Inclusion Criteria:

1. unresectable or recurrent GC histologically confirmed to be primary adenocarcinoma of the stomach.
2. age over 20 years.
3. Eastern Cooperative Oncology Group performance status score of 0-2.
4. written informed consent following full study information is provided to the patient.
5. progression or intolerance for first-line chemotherapy comprising fluorinated pyrimidine and platinum anticancer drugs (cisplatin or oxaliplatin) for advanced GC.
6. presence of evaluable lesions as confirmed using a computed tomography (CT) or magnetic resonance imaging.

Exclusion Criteria:

1. Patients with a life expectancy of shorter than 3 months
2. Patients with severe complications (angina pectoris, myocardial infarction, or arrhythmia) or uncontrollable diabetes mellitus, blood hypertension, or bleeding tendency.
3. Patients with a history of serious allergic reactions or serious drug allergy.
4. Patients with a clinically relevant mental disorder that prohibits response to questionnaires.
5. Patients for whom the attending physician considered that enrollment in the study is inappropriate.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients need second-line chemotherapy with unresectable or recurrent Gastric cancer.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Chemotherapy response | 2 years
  Follows by response valuation criteria in solid tumors (RECIST) evaluation. Partial response (PR) and Stable disease (SD) are defined as treatment effective, while Progressive disease (PD) is defined as no treatment effective.

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Takiguchi, PhD, Principal Investigator — City of Hope Medical Center
Locations (2):
- Department of Molecular Diagnostics and Experimental Therapeutics, Monrovia, California, United States
- Kawasaki Medical University, Kurashiki, Okayama-ken, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Ajani JA, D'Amico TA, Bentrem DJ, Chao J, Cooke D, Corvera C, Das P, Enzinger PC, Enzler T, Fanta P, Farjah F, Gerdes H, Gibson MK, Hochwald S, Hofstetter WL, Ilson DH, Keswani RN, Kim S, Kleinberg LR, Klempner SJ, Lacy J, Ly QP, Matkowskyj KA, McNamara M, Mulcahy MF, Outlaw D, Park H, Perry KA, Pimiento J, Poultsides GA, Reznik S, Roses RE, Strong VE, Su S, Wang HL, Wiesner G, Willett CG, Yakoub D, Yoon H, McMillian N, Pluchino LA. Gastric Cancer, Version 2.2022, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2022 Feb;20(2):167-192. doi: 10.6004/jnccn.2022.0008. PMID 35130500
- [Background] Fuchs CS, Tomasek J, Yong CJ, Dumitru F, Passalacqua R, Goswami C, Safran H, Dos Santos LV, Aprile G, Ferry DR, Melichar B, Tehfe M, Topuzov E, Zalcberg JR, Chau I, Campbell W, Sivanandan C, Pikiel J, Koshiji M, Hsu Y, Liepa AM, Gao L, Schwartz JD, Tabernero J; REGARD Trial Investigators. Ramucirumab monotherapy for previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (REGARD): an international, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2014 Jan 4;383(9911):31-39. doi: 10.1016/S0140-6736(13)61719-5. Epub 2013 Oct 3. PMID 24094768
- [Background] Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov O, Kim TY, Cunningham D, Rougier P, Komatsu Y, Ajani J, Emig M, Carlesi R, Ferry D, Chandrawansa K, Schwartz JD, Ohtsu A; RAINBOW Study Group. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1224-35. doi: 10.1016/S1470-2045(14)70420-6. Epub 2014 Sep 17. PMID 25240821
- [Background] Xu RH, Zhang Y, Pan H, Feng J, Zhang T, Liu T, Qin Y, Qin S, Yin X, Liu B, Ba Y, Yang N, Voon PJ, Tanasanvimon S, Zhou C, Zhang WL, Shen L. Efficacy and safety of weekly paclitaxel with or without ramucirumab as second-line therapy for the treatment of advanced gastric or gastroesophageal junction adenocarcinoma (RAINBOW-Asia): a randomised, multicentre, double-blind, phase 3 trial. Lancet Gastroenterol Hepatol. 2021 Dec;6(12):1015-1024. doi: 10.1016/S2468-1253(21)00313-7. Epub 2021 Oct 7. PMID 34626550
- [Background] Van Cutsem E, Muro K, Cunningham D, Bodoky G, Sobrero A, Cascinu S, Ajani J, Oh SC, Al-Batran SE, Wainberg ZA, Wijayawardana SR, Melemed S, Ferry D, Hozak RR, Ohtsu A; RAINBOW Investigators. Biomarker analyses of second-line ramucirumab in patients with advanced gastric cancer from RAINBOW, a global, randomized, double-blind, phase 3 study. Eur J Cancer. 2020 Mar;127:150-157. doi: 10.1016/j.ejca.2019.10.026. Epub 2020 Jan 31. PMID 32014812
- [Background] Natsume M, Shimura T, Iwasaki H, Okuda Y, Kitagawa M, Okamoto Y, Hayashi K, Kataoka H. Placental growth factor is a predictive biomarker for ramucirumab treatment in advanced gastric cancer. Cancer Chemother Pharmacol. 2019 Jun;83(6):1037-1046. doi: 10.1007/s00280-019-03817-2. Epub 2019 Mar 21. PMID 30899983
- [Background] Aprile G, Ongaro E, Del Re M, Lutrino SE, Bonotto M, Ferrari L, Rihawi K, Cardellino GG, Pella N, Danesi R, Fasola G. Angiogenic inhibitors in gastric cancers and gastroesophageal junction carcinomas: A critical insight. Crit Rev Oncol Hematol. 2015 Aug;95(2):165-78. doi: 10.1016/j.critrevonc.2015.02.009. Epub 2015 Mar 5. PMID 25800976
- [Background] Shigeyasu K, Toden S, Zumwalt TJ, Okugawa Y, Goel A. Emerging Role of MicroRNAs as Liquid Biopsy Biomarkers in Gastrointestinal Cancers. Clin Cancer Res. 2017 May 15;23(10):2391-2399. doi: 10.1158/1078-0432.CCR-16-1676. Epub 2017 Jan 31. PMID 28143873
- [Background] Yu W, Hurley J, Roberts D, Chakrabortty SK, Enderle D, Noerholm M, Breakefield XO, Skog JK. Exosome-based liquid biopsies in cancer: opportunities and challenges. Ann Oncol. 2021 Apr;32(4):466-477. doi: 10.1016/j.annonc.2021.01.074. Epub 2021 Feb 4. PMID 33548389
- [Background] Tang XH, Guo T, Gao XY, Wu XL, Xing XF, Ji JF, Li ZY. Exosome-derived noncoding RNAs in gastric cancer: functions and clinical applications. Mol Cancer. 2021 Jul 30;20(1):99. doi: 10.1186/s12943-021-01396-6. PMID 34330299
- [Background] Huang T, Song C, Zheng L, Xia L, Li Y, Zhou Y. The roles of extracellular vesicles in gastric cancer development, microenvironment, anti-cancer drug resistance, and therapy. Mol Cancer. 2019 Mar 30;18(1):62. doi: 10.1186/s12943-019-0967-5. PMID 30925929
- [Background] Kalluri R, LeBleu VS. The biology, function, and biomedical applications of exosomes. Science. 2020 Feb 7;367(6478):eaau6977. doi: 10.1126/science.aau6977. PMID 32029601
- [Background] Tanioka H, Nagasaka T, Uno F, Inoue M, Okita H, Katata Y, Kanzaki H, Kuramochi H, Satake H, Shindo Y, Doi A, Nasu J, Yamashita H, Yamaguchi Y. The relationship between peripheral neuropathy and efficacy in second-line chemotherapy for unresectable advanced gastric cancer: a prospective observational multicenter study protocol (IVY). BMC Cancer. 2019 Oct 11;19(1):941. doi: 10.1186/s12885-019-6163-6. PMID 31604467
- [Background] Shitara K, Takashima A, Fujitani K, Koeda K, Hara H, Nakayama N, Hironaka S, Nishikawa K, Makari Y, Amagai K, Ueda S, Yoshida K, Shimodaira H, Nishina T, Tsuda M, Kurokawa Y, Tamura T, Sasaki Y, Morita S, Koizumi W. Nab-paclitaxel versus solvent-based paclitaxel in patients with previously treated advanced gastric cancer (ABSOLUTE): an open-label, randomised, non-inferiority, phase 3 trial. Lancet Gastroenterol Hepatol. 2017 Apr;2(4):277-287. doi: 10.1016/S2468-1253(16)30219-9. Epub 2017 Jan 19. PMID 28404157
- [Background] Bando H, Shimodaira H, Fujitani K, Takashima A, Yamaguchi K, Nakayama N, Takahashi T, Oki E, Azuma M, Nishina T, Hironaka S, Komatsu Y, Shitara K. A phase II study of nab-paclitaxel in combination with ramucirumab in patients with previously treated advanced gastric cancer. Eur J Cancer. 2018 Mar;91:86-91. doi: 10.1016/j.ejca.2017.11.032. Epub 2018 Jan 30. PMID 29353164
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Fan Y, Siklenka K, Arora SK, Ribeiro P, Kimmins S, Xia J. miRNet - dissecting miRNA-target interactions and functional associations through network-based visual analysis. Nucleic Acids Res. 2016 Jul 8;44(W1):W135-41. doi: 10.1093/nar/gkw288. Epub 2016 Apr 21. PMID 27105848
- [Background] Joshi SS, Badgwell BD. Current treatment and recent progress in gastric cancer. CA Cancer J Clin. 2021 May;71(3):264-279. doi: 10.3322/caac.21657. Epub 2021 Feb 16. PMID 33592120
- [Background] Alsina M, Arrazubi V, Diez M, Tabernero J. Current developments in gastric cancer: from molecular profiling to treatment strategy. Nat Rev Gastroenterol Hepatol. 2023 Mar;20(3):155-170. doi: 10.1038/s41575-022-00703-w. Epub 2022 Nov 7. PMID 36344677
- [Background] Kang YK, Chen LT, Ryu MH, Oh DY, Oh SC, Chung HC, Lee KW, Omori T, Shitara K, Sakuramoto S, Chung IJ, Yamaguchi K, Kato K, Sym SJ, Kadowaki S, Tsuji K, Chen JS, Bai LY, Oh SY, Choda Y, Yasui H, Takeuchi K, Hirashima Y, Hagihara S, Boku N. Nivolumab plus chemotherapy versus placebo plus chemotherapy in patients with HER2-negative, untreated, unresectable advanced or recurrent gastric or gastro-oesophageal junction cancer (ATTRACTION-4): a randomised, multicentre, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2022 Feb;23(2):234-247. doi: 10.1016/S1470-2045(21)00692-6. Epub 2022 Jan 11. PMID 35030335
- [Background] Shitara K, Van Cutsem E, Bang YJ, Fuchs C, Wyrwicz L, Lee KW, Kudaba I, Garrido M, Chung HC, Lee J, Castro HR, Mansoor W, Braghiroli MI, Karaseva N, Caglevic C, Villanueva L, Goekkurt E, Satake H, Enzinger P, Alsina M, Benson A, Chao J, Ko AH, Wainberg ZA, Kher U, Shah S, Kang SP, Tabernero J. Efficacy and Safety of Pembrolizumab or Pembrolizumab Plus Chemotherapy vs Chemotherapy Alone for Patients With First-line, Advanced Gastric Cancer: The KEYNOTE-062 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020 Oct 1;6(10):1571-1580. doi: 10.1001/jamaoncol.2020.3370. PMID 32880601
- [Background] Hironaka S, Ueda S, Yasui H, Nishina T, Tsuda M, Tsumura T, Sugimoto N, Shimodaira H, Tokunaga S, Moriwaki T, Esaki T, Nagase M, Fujitani K, Yamaguchi K, Ura T, Hamamoto Y, Morita S, Okamoto I, Boku N, Hyodo I. Randomized, open-label, phase III study comparing irinotecan with paclitaxel in patients with advanced gastric cancer without severe peritoneal metastasis after failure of prior combination chemotherapy using fluoropyrimidine plus platinum: WJOG 4007 trial. J Clin Oncol. 2013 Dec 10;31(35):4438-44. doi: 10.1200/JCO.2012.48.5805. Epub 2013 Nov 4. PMID 24190112
- [Background] Shitara K, Doi T, Dvorkin M, Mansoor W, Arkenau HT, Prokharau A, Alsina M, Ghidini M, Faustino C, Gorbunova V, Zhavrid E, Nishikawa K, Hosokawa A, Yalcin S, Fujitani K, Beretta GD, Cutsem EV, Winkler RE, Makris L, Ilson DH, Tabernero J. Trifluridine/tipiracil versus placebo in patients with heavily pretreated metastatic gastric cancer (TAGS): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2018 Nov;19(11):1437-1448. doi: 10.1016/S1470-2045(18)30739-3. Epub 2018 Oct 21. PMID 30355453
- [Background] Shitara K, Bang YJ, Iwasa S, Sugimoto N, Ryu MH, Sakai D, Chung HC, Kawakami H, Yabusaki H, Lee J, Saito K, Kawaguchi Y, Kamio T, Kojima A, Sugihara M, Yamaguchi K; DESTINY-Gastric01 Investigators. Trastuzumab Deruxtecan in Previously Treated HER2-Positive Gastric Cancer. N Engl J Med. 2020 Jun 18;382(25):2419-2430. doi: 10.1056/NEJMoa2004413. Epub 2020 May 29. PMID 32469182
- [Background] Fornaro L, Musettini G, Orlandi P, Pecora I, Vivaldi C, Banchi M, Salani F, Fini E, Massa V, Catanese S, Cucchiara F, Lencioni M, Masi G, Vasile E, Bocci G. Early increase of plasma soluble VEGFR-2 is associated with clinical benefit from second-line treatment of paclitaxel and ramucirumab in advanced gastric cancer. Am J Cancer Res. 2022 Jul 15;12(7):3347-3356. eCollection 2022. PMID 35968330
- [Background] Sundar R, Barr Kumarakulasinghe N, Huak Chan Y, Yoshida K, Yoshikawa T, Miyagi Y, Rino Y, Masuda M, Guan J, Sakamoto J, Tanaka S, Tan AL, Hoppe MM, Jeyasekharan AD, Ng CCY, De Simone M, Grabsch HI, Lee J, Oshima T, Tsuburaya A, Tan P. Machine-learning model derived gene signature predictive of paclitaxel survival benefit in gastric cancer: results from the randomised phase III SAMIT trial. Gut. 2022 Apr;71(4):676-685. doi: 10.1136/gutjnl-2021-324060. Epub 2021 May 12. PMID 33980610
- [Background] Meng Q, Tan S, Jiang Y, Han J, Xi Q, Zhuang Q, Wu G. Post-discharge oral nutritional supplements with dietary advice in patients at nutritional risk after surgery for gastric cancer: A randomized clinical trial. Clin Nutr. 2021 Jan;40(1):40-46. doi: 10.1016/j.clnu.2020.04.043. Epub 2020 Jun 2. PMID 32563598
- [Background] Kawamura T, Makuuchi R, Tokunaga M, Tanizawa Y, Bando E, Yasui H, Aoyama T, Inano T, Terashima M. Long-Term Outcomes of Gastric Cancer Patients with Preoperative Sarcopenia. Ann Surg Oncol. 2018 Jun;25(6):1625-1632. doi: 10.1245/s10434-018-6452-3. Epub 2018 Apr 9. PMID 29633095
- [Background] Kamiya H, Komatsu S, Nishibeppu K, Ohashi T, Konishi H, Shiozaki A, Kubota T, Fujiwara H, Otsuji E. Obesity paradox as a new insight from postoperative complications in gastric cancer. Sci Rep. 2023 Jun 21;13(1):10116. doi: 10.1038/s41598-023-36968-7. PMID 37344511